CLINICAL TRIAL: NCT00002722
Title: RANDOMIZED PHASE II STUDY OF A WEEKLY 24H-INFUSION OF HIGH-DOSE 5-FU PLUS OR MINUS FOLINIC ACID (HD-FU/FA) VERSUS HD-FU/FA PLUS BIWEEKLY CISPLATIN VERSUS FAMTX (5-FU/ADRIAMYCIN/METHOTREXATE) IN ADVANCED GASTRIC CANCER, AN EORTC/AIO INTERGROUP TRIAL
Brief Title: High-Dose Chemotherapy in Treating Patients With Advanced Stomach Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: European Organisation for Research and Treatment of Cancer - EORTC (Network)
Responsible Party: Sponsor
Allocation: Randomized | Purpose: Treatment
Other Study IDs: EORTC-40953; EORTC-40953; GER-AIO-02/95
Record Dates: First submitted 1999-11-01; First posted 2004-04-22 (Estimated); Last update posted 2012-03-05 (Estimated); Status verified 2012-03

CONDITIONS: Gastric Cancer
Keywords: stage III gastric cancer; stage IV gastric cancer
MeSH Terms: conditions — Stomach Neoplasms | interventions — Cisplatin; Fluorouracil; Leucovorin

INTERVENTIONS:
Drug: cisplatin
Drug: fluorouracil
Drug: leucovorin calcium

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug and giving higher doses may kill more tumor cells.

PURPOSE: Randomized phase II trial to study the effectiveness of high-dose chemotherapy in treating patients with advanced stomach cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the response rates in patients with advanced gastric cancer treated with high-dose fluorouracil (5-FU) with vs without high-dose leucovorin (CF) vs high-dose 5-FU/CF/cisplatin. II. Determine the toxic effects of these regimens in these patients. III. Assess the symptomatic improvement in these patients treated with these regimens.

OUTLINE: This is a randomized, multicenter study. Patients are stratified according to participating center, WHO performance status (0 or 1 vs 2), and disease stage (metastatic vs locally advanced). Patients are randomized to 1 of 3 treatment arms. Arm I: Patients receive fluorouracil (5-FU) IV over 24 hours weekly for 6 weeks. Arm II: Patients receive leucovorin calcium (CF) IV over 2 hours followed by 5-FU IV over 24 hours weekly for 6 weeks. Arm III: Patients receive CF and 5-FU as in arm II and cisplatin IV over 1 hour on days 1, 15, and 29. Treatment repeats every 7 weeks for a maximum of 4 courses in the absence of unacceptable toxicity or disease progression. Patients are followed every 8 weeks.

PROJECTED ACCRUAL: A total of 65-135 patients (21-45 per arm) will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed gastric cancer that is either metastatic or locally advanced and inoperable Bidimensionally measurable disease No CNS metastasis

PATIENT CHARACTERISTICS: Age: 75 and under Performance status: WHO 0-2 Life expectancy: At least 3 months Hematopoietic: Granulocyte count at least 2,000/mm3 Platelet count at least 100,000/mm3 Hepatic: Bilirubin no greater than 1.7 mg/dL Renal: Creatinine no greater than 1.3 mg/dL Creatinine clearance greater than 60 mL/min Cardiovascular: No myocardial infarction within past 12 months No coronary heart disease requiring drug therapy Congestive heart failure or arrhythmia treatable with standard medication allowed Other: No active infection No history of severe mental disorder No other malignancy within past 10 years except carcinoma in situ of the cervix or nonmelanoma skin cancer Not pregnant

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: No prior chemotherapy Endocrine therapy: Not specified Radiotherapy: No prior radiotherapy Surgery: Not specified

Max Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 135 (Estimated)
Dates: Start 1996-01; Primary Completion 1999-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hansjochen Wilke, MD, Study Chair — Kliniken Essen-Mitte